CLINICAL TRIAL: NCT05718310
Title: Habituation of the Nociceptive Blink Reflex in Experimentally Induced Migraine Attack: a Cross-over, Randomized Controlled Study
Brief Title: Habituation of the Nociceptive Blink Reflex in Experimentally Induced Migraine Attack
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Collaborators: University of Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: NTG_nBR
Record Dates: First submitted 2023-01-19; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Migraine; Migraine Disorders; Pain
MeSH Terms: conditions — Migraine Disorders; Pain | interventions — Nitroglycerin; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitroglycerin (Active Comparator): Nitroglycerin diluted in 250 ml of sodium chloride 0.9% will be administered once via an infusion pump intravenously, at a dose of 0.5 μg/kg/min in 20 minutes.
  Interventions: Drug: Nitroglycerin
- Saline (Placebo Comparator): 250 ml of sodium chloride 0.9% will be administered intravenously in 20 minutes via an infusion pump.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Nitroglycerin — 25 migraine patients without aura of both genders are randomized to receive a 20-minutes infusion of NTG and/or sterile saline on two days, with at least one week in between
  Other Names: NTG
  Arms: Nitroglycerin
Drug: Saline — 25 migraine patients without aura of both genders are randomized to receive a 20-minutes infusion of NTG and/or sterile saline on two days, with at least one week in between
  Other Names: Isotonic saline; 0.9% NaCl
  Arms: Saline

SUMMARY:
People with migraine typically show impaired responsivity to visual, auditory and pain stimuli (Burstein et al, 2015). The electrophysiological study of the nociceptive blink reflex (nBR) is widely adopted for the instrumental evaluation of trigeminal afferent function.

Migraine sufferers characteristically show deficits in the habituation to repeated stimulations of various sensory modalities, in the interictal phase of the disease (Bohotin et al, 2002; Di Clemente et al, 2005).

It has been described how the habituation / sensitization pattern presents a characteristic pattern over the course of the migraine cycle. Past evidence suggests that the habituation deficit may turn towards a normalization of the pattern near the acute migraine attack (Coppola et al, 2013; Katsarava et al, 2003).

However, the study of the spontaneous attack shows various limits and difficulties, mainly due to the impossibility of predicting the onset of the next attack and of standardizing the experimental conditions. The use of human models of migraine allows us to overcome these obstacles. Di Clemente et al. (2009) evaluated the electrophysiological changes in nBR after administration of nitroglycerin (NTG) in healthy subjects. The authors described a modification of trigeminal circuits and cortical responses (visual evoked potentials) after NTG. However, NTG administration does not induce migraine attack in healthy subjects, therefore this model cannot be directly translated to migraine pathology (Ashina et al. 2017).

Our group has previously used the human model of migraine based on the administration of NTG to study central and spinal level sensitization through the nociceptive avoidance reflex in the lower limb (RIII) (De Icco et al. 2020). The results of the previous study deepened our understanding of the central mechanisms of sensitization.

The investigation of the nBR allows to study the modulation of the caudal trigeminal complex (TCC). In the present study we therefore intend to evaluate, under well-controlled experimental conditions, the modulation of the trigeminal caudal complex during an experimentally induced migraine attack. The study will allow us to confirm or not the normalization of habituation described in the acute phase through the adoption of a solid cross-over and placebo-controlled study design.

DETAILED DESCRIPTION:
This is an interventional, randomized, crossover and double-blind placebo-controlled study. The enrolled subjects will participate in two study sessions (V1 and V2, respectively) placed at least one week apart.

A first screening visit (V0) is planned, during which the clinical-demographic data will be collected, the patients will undergo a complete neurological and objective examination, and an ECG will be performed to exclude major cardiac pathologies. Patients who meet the inclusion / exclusion criteria will continue with the subsequent study sessions (V1 and V2). During V1 and V2 the subjects must be in the inter-critical phase of the disease, i.e. free from headache and in the absence of analgesic drugs in the previous 48 hours.

First study session (V1):

At baseline (T0), disease assessment scales (MIDAS, HIT-6, ASC-12, MSQ, BDI, STAI) will be administered, and the first electrophysiological test session (nociceptive blink reflex -nBR) will be performed along with the first blood sample from a peripheral venous catheter positioned in the antecubital vein.

At the end of the baseline evaluation, the subjects will be randomized into two groups to receive, during the first of the two sessions, NTG (0.5 μg / kg / min intravenous in 20 minutes) or placebo (intravenous saline in 20 minutes) via infusion pump.

The subjects will then be monitored in hospital for 4 hours following the NTG infusion (hospital phase) and then discharged with the indication to keep a headache diary for a further 8 hours (12 hours of overall observation). At the end of the 4 hours of hospital observation, the investigator or the patient may decide to extend the observation period based on the possible occurrence of adverse effects or in any case as required.

Starting from the infusion, the onset of headache and associated characteristics (nausea, vomiting, photophobia, phonophobia, location of pain, quality of pain, aggravation with cough, intensity) will be evaluated every ten minutes, as well as the presence of other symptoms or adverse events. The vital parameters (blood pressure, heart rate) will be monitored every 5 minutes during the infusion, then every 10 minutes for the entire duration of the in-hospital observation. Additional vital sign measurements will be performed based on clinical need or trend.

After 2 hours (T1) and 4 hours (T2) from the end of the NTG / placebo infusion, the electrophysiological evaluations and blood samples will be repeated, and the assessment scale for allodynia (ASC-12) will be administered.

In subjects in which the induced migraine attack will appear within the hospital observation phase (4 hours), sumatriptan 6 mg will be administered subcutaneously. 1 hour after the administration of sumatriptan, the electrophysiological evaluation of the nBR and blood sampling after (TS) will be repeated.

Second study session (V2):

Patients will return to the center for the second session (V2) of the study at least one week after the first session. The second session will completely mirror the first, patients will receive placebo (intravenous saline in 20 minutes) or NTG (0.5 μg / kg / min intravenous in 20 minutes) in cross-over according to the randomization list.

It is specified that, for female subjects, a urine pregnancy test will be carried out before each study session.

The patient will be informed that headache may arise during the test, but no information will be shared on the possible course after NTG / placebo to avoid breaking the blind.

NBR registration procedure:

The R2 response of nBR will be evaluated using a planar concentric electrode (Bionen, Florence, Italy), placed 10 mm above the emergence of the supraorbital nerve. For each subject, the preferential side of pain localization of migraine crises will be chosen, alternatively the right side will be used. Stimulation parameters: single monopolar stimulation, duration 0.3 ms, band filter: 3 Hz to 3 kHz, recording frequency: 2.5 kHz, analysis time: 200ms, sensitivity: 100 mV.

The surface electromyographic recording (CED Powerlab 1401, Cambridge Electronic Design) will be carried out at the level of the orbicularis oculi muscle through a pair of surface electrodes, the reference electrode on the side of the eye, the recording electrode on the midpoint of the lower eyelid. A progressive increase in the stimulation intensity (0.3 mA at a time) will be used to evaluate the reflex threshold (RT = reflex threshold), defined as a stably present response to at least 3 stimulations. To assess the habituation of nBR, 26 consecutive stimuli will be administered at different stimulus frequencies, according to a random order (0.2, 0.3, 0.5 Hz), with a stimulation intensity equal to 1.8 times the RT. Of these stimulations, the first will be removed from the analysis to eliminate the startle response. The 25 electromyographic recordings will be collected in 5 blocks, and the values of the area under the amplitude curve (AUC, ms * mV) will be calculated for each block. The percentage change in the AUC of the last block, compared to the first, represents the "habituation index" (HI) value.

Biochemical panel:

* Plasma levels of pro and anti inflammatory cytokines (TNF-alpha, IL-1beta, IL-6, IL-4, IL-10) through a latest generation ELISA analysis
* Plasma levels of quinolinic acid, through mass spectrometry;
* Plasma levels of CGRP, PACAP, VIP through commercially available ELISA kits.
* Gene expression of the cytokines mentioned above and specific microRNAs (mir-155, mir-382, mir-34a, mir-30a) and MALAT1 through RT-PCR method.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of "1.1 Migraine without aura", according to ICHD-3 criteria, with a history of disease of at least one year;
* Frequency between 3 and 14 migraine days per month;
* Have completed a prospective headache diary for at least 1 month to confirm diagnosis and frequency.

Exclusion Criteria:

* Current or previous diagnosis of other forms of primary or secondary headache according to ICHD-3 criteria; it will be possible to enroll patients diagnosed with "2.1 Sporadic episodic tension-type headache", according to ICHD-3 criteria;
* Other conditions causing chronic pain;
* Significant cardiovascular disorders;
* History of other neurological or psychiatric disorders that may affect the study assessments;
* Contraindications or intolerance to the administration of Sumatriptan or NTG;
* Use of more than 1 preventive drug for the treatment of migraine, according to national guidelines;
* Change in the dosage of prevention treatment for migraine in the last month;
* Women in current or planned pregnancy, and breastfeeding;
* Chronic use of active ingredients with analgesic or sedative action (steroids, opioids, anti-inflammatories, paracetamol) or in any case capable of modifying the pain threshold (for example tricyclic antidepressants or serotonin reuptake inhibitors);
* Use of phosphodiesterase inhibitors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Difference in the habituation index between the experimental and control group | Change from baseline (T0) to 2 hours after infusion (T1) to 4 hours after infusion (T2)
  The primary outcome is to assess the difference of the habituation index between the NTG exposed group and the placebo group across the main timepoints

SECONDARY OUTCOMES:
Difference in the habituation index in the experimental group treated with sumatriptan | Change from baseline (T0) to 2 hours after infusion (T1) to 4 hours after infusion (T2) to 1 hour after sumatriptan injection (TS)
  A secondary outcome is the difference of the habituation index in patients exposed to NTG who will develop headache with migraine features during the in-hospital observation period, and will be subsequently treated with sumatriptan, as compared to the remaining timepoints
Difference in the nociceptive blink reflex threshold between the experimental and control group | Change from baseline (T0) to 2 hours after infusion (T1) to 4 hours after infusion (T2)
  A secondary outcome is to assess the difference of the nociceptive blink reflex threshold between the NTG exposed group and the placebo group across the main timepoints
Difference in the nociceptive blink reflex threshold in the experimental group treated with sumatriptan | Change from baseline (T0) to 2 hours after infusion (T1) to 4 hours after infusion (T2) to 1 hour after sumatriptan injection (TS)
  A secondary outcome is to assess the difference of the nociceptive blink reflex threshold in patients exposed to NTG who will develop headache with migraine features during the in-hospital observation period, and will be subsequently treated with sumatriptan, as compared to the remaining timepoints
Difference in the inflammatory cytokines expression between the experimental and control group | Change from baseline (T0) to 2 hours after infusion (T1) to 4 hours after infusion (T2)
  A secondary outcome is the difference of TNF-alpha, IL-1beta, IL-6, IL-4, IL-10 plasma levels between the NTG exposed group and the placebo group across the main timepoints
Difference in the inflammatory cytokines expression in the in the experimental group treated with sumatriptan | Change from baseline (T0) to 2 hours after infusion (T1) to 4 hours after infusion (T2) to 1 hour after sumatriptan injection (TS)
  A secondary outcome is the difference of TNF-alpha, IL-1beta, IL-6, IL-4, IL-10 plasma levels in patients exposed to NTG who will develop headache with migraine features during the in-hospital observation period, and will be subsequently treated with sumatriptan, as compared to the remaining timepoints
Difference in the quinolinic acid panel expression between the experimental and control group | Change from baseline (T0) to 2 hours after infusion (T1) to 4 hours after infusion (T2)
  A secondary outcome is the difference of quinolinic acid plasma levels between the NTG exposed group and the placebo group across the main timepoints
Difference in the quinolinic acid panel expression between in the experimental group treated with sumatriptan | Change from baseline (T0) to 2 hours after infusion (T1) to 4 hours after infusion (T2) to 1 hour after sumatriptan injection (TS)
  A secondary outcome is the difference of quinolinic acid plasma levels in patients exposed to NTG who will develop headache with migraine features during the in-hospital observation period, and will be subsequently treated with sumatriptan, as compared to the remaining timepoints
Difference in the CGRP expression between the experimental and control group | Change from baseline (T0) to 2 hours after infusion (T1) to 4 hours after infusion (T2)
  A secondary outcome is the difference of CGRP plasma levels between the NTG exposed group and the placebo group across the main timepoints
Difference in the PACAP expression between the experimental and control group | Change from baseline (T0) to 2 hours after infusion (T1) to 4 hours after infusion (T2)
  A secondary outcome is the difference of PACAP plasma levels between the NTG exposed group and the placebo group across the main timepoints
Difference in the VIP expression between the experimental and control group | Change from baseline (T0) to 2 hours after infusion (T1) to 4 hours after infusion (T2)
  A secondary outcome is the difference of VIP plasma levels between the NTG exposed group and the placebo group across the main timepoints
Difference in the CGRP expression in the experimental group treated with sumatriptan | Change from baseline (T0) to 2 hours after infusion (T1) to 4 hours after infusion (T2) to 1 hour after sumatriptan injection (TS)
  A secondary outcome is the difference of CGRP plasma levels in patients exposed to NTG who will develop headache with migraine features during the in-hospital observation period, and will be subsequently treated with sumatriptan, as compared to the remaining timepoints
Difference in the PACAP expression in the experimental group treated with sumatriptan | Change from baseline (T0) to 2 hours after infusion (T1) to 4 hours after infusion (T2) to 1 hour after sumatriptan injection (TS)
  A secondary outcome is the difference of PACAP plasma levels in patients exposed to NTG who will develop headache with migraine features during the in-hospital observation period, and will be subsequently treated with sumatriptan, as compared to the remaining timepoints
Difference in the VIP expression in the experimental group treated with sumatriptan | Change from baseline (T0) to 2 hours after infusion (T1) to 4 hours after infusion (T2) to 1 hour after sumatriptan injection (TS)
  A secondary outcome is the difference of VIP plasma levels in patients exposed to NTG who will develop headache with migraine features during the in-hospital observation period, and will be subsequently treated with sumatriptan, as compared to the remaining timepoints
Difference in the epigenetic panel expression between the experimental and control group | Change from baseline (T0) to 2 hours after infusion (T1) to 4 hours after infusion (T2)
  A secondary outcome is the difference of mir-155, mir-382, mir-34a, mir-30a, MALAT1 plasma levels between the NTG exposed group and the placebo group across the main timepoints
Difference in the epigenetic panel expression in the experimental group treated with sumatriptan | Change from baseline (T0) to 2 hours after infusion (T1) to 4 hours after infusion (T2) to 1 hour after sumatriptan injection (TS)
  A secondary outcome is the difference of mir-155, mir-382, mir-34a, mir-30a, MALAT1 plasma levels in patients exposed to NTG who will develop headache with migraine features during the in-hospital observation period, and will be subsequently treated with sumatriptan, as compared to the remaining timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Roberto De Icco, MD, Principal Investigator — IRCCS, Mondino Foundation
Locations (2):
- Italy (2):
  - Headache Science & Neurorehabilitation Center, Pavia
  - IRCCS Mondino Foundation, Pavia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burstein R, Noseda R, Borsook D. Migraine: multiple processes, complex pathophysiology. J Neurosci. 2015 Apr 29;35(17):6619-29. doi: 10.1523/JNEUROSCI.0373-15.2015. PMID 25926442
- [Background] Bohotin V, Fumal A, Vandenheede M, Gerard P, Bohotin C, Maertens de Noordhout A, Schoenen J. Effects of repetitive transcranial magnetic stimulation on visual evoked potentials in migraine. Brain. 2002 Apr;125(Pt 4):912-22. doi: 10.1093/brain/awf081. PMID 11912123
- [Background] Di Clemente L, Coppola G, Magis D, Fumal A, De Pasqua V, Schoenen J. Nociceptive blink reflex and visual evoked potential habituations are correlated in migraine. Headache. 2005 Nov-Dec;45(10):1388-93. doi: 10.1111/j.1526-4610.2005.00271.x. PMID 16324171
- [Background] Coppola G, Di Lorenzo C, Schoenen J, Pierelli F. Habituation and sensitization in primary headaches. J Headache Pain. 2013 Jul 30;14(1):65. doi: 10.1186/1129-2377-14-65. PMID 23899115
- [Background] Di Clemente L, Coppola G, Magis D, Gerardy PY, Fumal A, De Pasqua V, Di Piero V, Schoenen J. Nitroglycerin sensitises in healthy subjects CNS structures involved in migraine pathophysiology: evidence from a study of nociceptive blink reflexes and visual evoked potentials. Pain. 2009 Jul;144(1-2):156-61. doi: 10.1016/j.pain.2009.04.018. Epub 2009 May 19. PMID 19457613
- [Background] Ashina M, Hansen JM, A Dunga BO, Olesen J. Human models of migraine - short-term pain for long-term gain. Nat Rev Neurol. 2017 Dec;13(12):713-724. doi: 10.1038/nrneurol.2017.137. Epub 2017 Oct 6. PMID 28984313
- [Background] De Icco R, Perrotta A, Grillo V, Cosentino G, Sances G, Sandrini G, Tassorelli C. Experimentally induced spinal nociceptive sensitization increases with migraine frequency: a single-blind controlled study. Pain. 2020 Feb;161(2):429-438. doi: 10.1097/j.pain.0000000000001726. PMID 31633594
- [Background] Sances G, Tassorelli C, Pucci E, Ghiotto N, Sandrini G, Nappi G. Reliability of the nitroglycerin provocative test in the diagnosis of neurovascular headaches. Cephalalgia. 2004 Feb;24(2):110-9. doi: 10.1111/j.1468-2982.2004.00639.x. PMID 14728706
- [Background] De Icco R, Greco R, Demartini C, Vergobbi P, Zanaboni A, Tumelero E, Reggiani A, Realini N, Sances G, Grillo V, Allena M, Tassorelli C. Spinal nociceptive sensitization and plasma palmitoylethanolamide levels during experimentally induced migraine attacks. Pain. 2021 Sep 1;162(9):2376-2385. doi: 10.1097/j.pain.0000000000002223. PMID 33587406
- [Background] Karsan N, Perez-Rodriguez A, Nagaraj K, Bose PR, Goadsby PJ. The migraine postdrome: Spontaneous and triggered phenotypes. Cephalalgia. 2021 May;41(6):721-730. doi: 10.1177/0333102420975401. Epub 2021 Jan 10. PMID 33423506
- [Background] Demartini C, Greco R, Zanaboni AM, Sances G, De Icco R, Borsook D, Tassorelli C. Nitroglycerin as a comparative experimental model of migraine pain: From animal to human and back. Prog Neurobiol. 2019 Jun;177:15-32. doi: 10.1016/j.pneurobio.2019.02.002. Epub 2019 Feb 13. PMID 30771365